CLINICAL TRIAL: NCT04799912
Title: Labor Induction in Low-risk Nulliparous Women at 39 Weeks of Gestation to Reduce Cesarean: A Randomized Trial of Induction Versus Expectant Management in France (FRENCH-ARRIVE)
Acronym: FRENCH-ARRIVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHUBX 2019/58
Record Dates: First submitted 2021-03-12; First posted 2021-03-16 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Cesarean Section
Keywords: Cesarean section; Labor induction; Expectant management; Low risk nulliparous women; Maternal morbidity; Neonatal morbidity

STUDY DESIGN:
Intervention Model Description: Multicenter open randomized controlled trial with 2 parallel arms
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elective labor induction (Experimental): Elective labor induction via oxytocin between 39 weeks of gestation and 0 day and 39 weeks of gestation and 4 days for women with favorable cervix. Those with an unfavorable cervix (Bishop score < 6) will first undergo cervical ripening (method left to the discretion of the practitioner) in conjunction with or followed by oxytocin stimulation unless a contraindication arises. Except for elective induction of labor between 39 weeks of gestation and 0 day and 39 weeks of gestation and 4 days, the obstetrical management will not be modified compared to routine obstetrical management.
  Interventions: Procedure: Elective labor induction
- Expectant management (No Intervention): Standard follow-up visits until at least 41 weeks of gestation and 0 day without elective labor induction unless a medical indication is present. Antepartum fetal testing will be initiated no later than 41 weeks of gestation and 1 day according to policies at each center (according to the French guidelines). If still pregnant, all women will undergo induction since 41 weeks of gestation but no later than 42 weeks of gestation (according to the French guidelines)

INTERVENTIONS:
Procedure: Elective labor induction — Elective labor induction at 39 weeks of gestation
  Arms: Elective labor induction

SUMMARY:
The recent ARRIVE trial conducted in United States of America in 2014-2017 demonstrates that elective induction of labor at 39 weeks for nulliparous women did result in a significantly lower frequency of cesarean delivery with no significant differences of adverse perinatal outcomes. But the expected benefits of elective labor induction at 39 weeks have to be confirmed in other settings outside US before considering routine induction of labor for all low-risk nulliparous women at 39 weeks of gestation worldwide.

DETAILED DESCRIPTION:
The nadir of the neonatal risks seems to be at 39 weeks of gestation and there is an augmentation of maternal complications after 39 weeks. Nonetheless, planned induction of labor at 39 weeks was not encouraged in common practice due to a suspected higher risk of frequency cesarean delivery and other adverse maternal outcomes, especially among nulliparous women with unfavorable cervix, compared with expectant management. This suspected increased maternal morbidity especially the cesarean rate associated with the induction of labor was based on observational studies which suffer from methodological limitations or based on underpowered small randomized clinical trials.

A recent multicenter, randomized, controlled, unmasked trial conducted in United States of America in 2014-2017 (ARRIVE trial), provides new results with a high level of evidence. This trial conducted among 6,106 low-risk nulliparous women who were randomized, 3062 assigned to labor induction at 39 weeks 0 day to 39 weeks 4 days and 3,044 assigned to expectant management, demonstrates that induction of labor at 39 weeks did result in a trend but not significant lower frequency of the primary outcome - a composite adverse perinatal outcome - (relative risk [RR] 0.80, 95% confidence interval [CI] 0.64-1.00), but did result in a significantly lower frequency of cesarean delivery (RR 0.84, 95% CI 0.76-0.93).

Although the cesarean delivery rate was a secondary outcome of the study and the absence of any comparison for women's characteristics of those who were eligible and declined to participate and those who were randomized, the recommendations of the Society of Maternal-Fetal Medicine (SMFM), American College of Obstetricians and Gynecologists (ACOG) and numerous authors have already considered that induction of labor ≥ 39 weeks should be proposed in low-risk nulliparous women. In other words, on the basis mainly on the results of a secondary outcome from only one single randomized controlled trial, they have proposed to modify the management of the pregnant women who reach 39 weeks gestation (i.e. the large majority of the pregnant women) while until now induction of labor for those women was proposed only if abnormal medical condition occurred or beyond 41 weeks of gestation. Nevertheless, the findings of the ARRIVE trial are so important because the reduction of the cesarean rate is a worldwide goal and the elective induction of labor ≥ 39 weeks seems to be today the most effective way to achieve it. However, French context and obstetrical practices are different than USA, with a lower rate of cesarean. Women's characteristics are also different (i.e. lower body mass index in France). Consequently, the external validity of the ARRIVE trial needs to be confirmed. Moreover, in the ARRIVE trial, the labor management has to respect American recent guidelines with a longer duration of the latent phase and administration of oxytocin if needed for at least 12 hours after membrane rupture before deeming the induction a failure. A generalization of labor induction at 39 weeks without a strictly respect of the eligibility criteria or labor management could result to an increase of unexpected adverse maternal or neonatal outcomes.

Thus, the expected benefits of labor induction at 39 weeks have to be confirmed in other context, in particular in French settings with a lower cesarean rate than in USA by replicating the ARRIVE study conducting another randomized controlled trial for which the primary outcome will be the cesarean section rate.

This replication is crucial before leading to a such important change in daily practice that would be considering routine induction of labor for low-risk nulliparous women at 39 weeks of gestation and consequently modifying the organization of all maternity wards in order to achieve this policy.

In addition to the replication of the ARRIVE trial in a French context, a prospective observational cohort with 4,200 women is associated with this trial to identify a potential participant selection bias.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Nulliparous women (i.e. no previous pregnancy beyond 20 weeks)
* With singleton gestation. Twin gestation reduced to singleton, either spontaneously or therapeutically, is not eligible unless the reduction occurred before 14 weeks project gestational age
* Gestational age at randomization between 37 weeks of gestation 0 day and 38 weeks of gestation 6 days inclusive based on the crown rump length measured at the first trimester ultrasound before 14 weeks of gestation and 0 day, as recommended in France
* Affiliated or beneficiary to a health security system
* Signed informed consent

Exclusion Criteria:

* Project gestational age at date of first ultrasound > 14 weeks
* Plan for induction of labor prior to 40 weeks 5 days
* Plan for cesarean delivery or contraindication to labor
* Breech presentation
* Multiple pregnancy
* Signs of labor (regular painful contractions with cervical change)
* Fetal demise or known major fetal anomaly
* Heparin or low-molecular weight heparin during the current pregnancy
* Placenta previa, accreta, vasa previa
* Active vaginal bleeding greater than bloody show
* Ruptured membranes
* Cerclage in current pregnancy
* Known oligohydramnios, defined as Amniotic Fluid Index < 5 or Maximal Vertical Pocket < 2 cm
* Fetal growth restriction, defined as Estimated Fetal Weight < 10th percentile according to local curve
* Known HIV positivity because of modified delivery plan
* Major maternal medical illness associated with increased risk for adverse pregnancy outcome (for example, any diabetes mellitus, lupus, any hypertensive disorder, cardiac disease, renal insufficiency)
* Refusal of blood products
* Contraindication to oxytocin
* Participation in another interventional study that influences management of labor or delivery (labor induction, operative vaginal delivery, cesarean section, shoulder dystocia)
* Delivery planned elsewhere at a non-Network site
* History of myomectomy by laparotomy or laparoscopy
* Previous metroplasty for uterine malformation or Asherman syndrome
* Patient under legal protection
* Poor understanding of the French language

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4200 (Estimated)
Dates: Start 2021-04-12 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of cesarean section | Day 1
  Incidence of cesarean section defined as a cesarean birth regardless of the indication from the time the woman is randomized

SECONDARY OUTCOMES:
Incidence of incisional extensions | Day 1
  Incidence of incisional extensions at cesarean section or cervical traumas
Incidence of operative vaginal delivery | Day 1
  Incidence of operative vaginal delivery and indication
Incidence of operative vaginal delivery for cesarean | Day 1
  Incidence of operative delivery defined by a cesarean delivery or an instrumental vaginal delivery
Incidence of third or fourth degree perineal laceration | Day 1
  Incidence of third or fourth degree perineal laceration
Incidence of chorioamnionitis | Hospital discharge (Day 3-5)
  Incidence of chorioamnionitis, defined as a clinical diagnosis before delivery as: maternal fever (body temperature ≥ 38°C) with no alternative cause identified and at least one sign among the following: fetal tachycardia>160 bpm for ≥ 10min or purulent amniotic fluid from the cervical canal
Incidence of postpartum hemorrhage | Hospital discharge (Day 3-5)
  Incidence of postpartum hemorrhage defined similarly as Grobman et al. in ARRIVE trial as any of the following:
  * Transfusion
  * Non-elective hysterectomy
  * Use of sulprostone
  * Other surgical interventions such as uterine compression sutures, uterine artery ligation, embolization and hypogastric ligation, balloon tamponade
  * Curettage
Incidence of admission to intensive care unit | Hospital discharge (Day 3-5)
  Incidence of admission to intensive care unit
Incidence of maternal death | Hospital discharge (Day 3-5)
  Incidence of maternal death
Incidence of preeclampsia/gestational hypertension | Hospital discharge (Day 3-5)
  Incidence of preeclampsia/gestational hypertension
Maternal pain | Hospital discharge (Day 3-5)
  Median patient-reported pain outcomes with a 10-point Likert scale
Maternal satisfaction | Hospital discharge (Day 3-5)
  Maternal satisfaction with a satisfaction questionnaire derived from the childbirth experience questionnaire and satisfaction questionnaire
interval from randomization to delivery | Day 1
  Median interval from randomization to delivery
gestational age at delivery | Day 1
  Median gestational age at delivery
Incidence of maternal postpartum infection | Hospital discharge (Day 3-5)
  Incidence of maternal postpartum infection defined similarly as Grobman et al. in ARRIVE trial as any of the following:
  * Clinical diagnosis of endometritis
  * Wound reopened for hematoma, seroma, infection or other reasons
  * Cellulitis requiring antibiotics
  * Pneumonia
  * Pyelonephritis
  * Bacteremia unknown source
  * Septic pelvic thrombosis
Incidence of maternal venous thromboembolism | Hospital discharge (Day 3-5)
  Incidence of maternal venous thromboembolism (deep venous thrombosis diagnosed using bilateral leg Doppler ultrasound or pulmonary embolism diagnosed using bilateral ventilation-perfusion lung scanning or computed tomographic pulmonary angiography)
Cervical ripening and induction | Day 1-2
  Method used for cervical ripening and induction
Incidence of composite of severe neonatal morbidity and perinatal mortality | Hospital discharge (Day 3-5)
  Incidence of composite of severe neonatal morbidity and perinatal mortality (any one of the following):
  * Antepartum, intrapartum, or neonatal death
  * Intubation, continuous positive airway pressure (CPAP) or high-flow nasal cannula (HFNC) for ventilation or cardiorespiratory support within first 72 hours
  * Apgar ≤ 3 at 5 minutes
  * Neonatal encephalopathy
  * Seizures
  * Sepsis (presence of a clinically ill infant in whom systemic infection is suspected with a positive blood, cerebral spinal fluid (CSF), or catheterized/suprapubic urine culture; or, in the absence of positive cultures, clinical evidence of cardiovascular collapse or an unequivocal X-ray confirming infection).
  * Pneumonia confirmed by X-ray or positive blood culture.
  * Meconium aspiration syndrome
  * Birth trauma (bone fractures, brachial plexus palsy, other neurologic injury, retinal hemorrhage, facial nerve injury)
  * Intracranial hemorrhage or subgaleal hemorrhage
  * Hypotension requiring pressor support
Mean birth weight | Day 1
  Mean birth weight, incidence of macrosomia > 4,000 g, incidence of large for date fetuses defined as > 90th percentile weight for gestational age
Incidence of neonatal acidosis | Day 1
  Incidence of neonatal acidosis (defined by umbilical cord arterial pH < 7.00)
Median duration of respiratory support | Hospital discharge (Day 3-5)
  Median duration of respiratory support including ventilator, CPAP, HFNC
Incidence of small for gestational age | Day 1
  Incidence of small for gestational age defined as < 5th and < 10th percentile weight for gestational age
Incidence of cephalohematoma | Hospital discharge (Day 3-5)
  Incidence of cephalohematoma
Incidence of shoulder dystocia | Day 1
  Incidence of shoulder dystocia
Incidence of neonatal transfusion | Hospital discharge (Day 3-5)
  Incidence of neonatal transfusion of blood products or blood
Incidence of hyperbilirubinemia | Hospital discharge (Day 3-5)
  Incidence of hyperbilirubinemia requiring phototherapy or exchange transfusion
Incidence of hypoglycemia | Hospital discharge (Day 3-5)
  Incidence of hypoglycemia (glucose < 35 mg/L) requiring IV therapy
Incidence of admission to neonatal intensive care unit | Hospital discharge (Day 3-5)
  Incidence of admission to neonatal intensive care unit or intermediate care unit
Incidence of epidural use | Day 1
  outcomes: Incidence of epidural use
Median hours on the labor and delivery unit | Day 1-2
  Median hours on the labor and delivery unit
Median maternal postpartum length of hospital stay | Hospital discharge (Day 3-5)
  Median maternal postpartum length of hospital stay
Median neonatal length of hospital stay | Hospital discharge (Day 3-5)
  Median neonatal length of hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: Undecided